CLINICAL TRIAL: NCT04112420
Title: Detection of the Incidence of Intensively Medically Relevant Pre-existing Cardio-pulmonary Diseases by Using of Focused Echocardiography Upon Admission to the Intensive Care Unit
Brief Title: Detection of the Incidence of Pre-existing Cardio-pulmonary Diseases by Using of Echocardiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Kilany, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FATE
Record Dates: First submitted 2019-09-25; First posted 2019-10-02 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2019-09

CONDITIONS: Intensive Care Unit Syndrome

STUDY DESIGN:
Intervention Model Description: 200 patients > 60 years with unplanned admission to the intensive care unit are to be included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group A (Other): 200 Participants more than 60 yrs old having Trans-esophageal Echocardiography examination upon admission to ICU
  Interventions: Diagnostic Test: Trans-esophageal echocardiography

INTERVENTIONS:
Diagnostic Test: Trans-esophageal echocardiography — The department registers an unplanned admission of a patient to the intensive care unit. The indication is verified again by the intensive care physician.
  In this case, the patient is then admitted to the intensive care unit, supervised by an intensive care physician, orientated and initiated therapeutic and diagnostic measures.
  As part of the planned transthoracic cardiac ultrasound examination, it is then selected whether the patient is suitable according to the patient's will and the inclusion or exclusion criteria.
  After clarification, time to think and consent, the examination is then carried out according to the protocol by approved doctors of the Clinic for Anesthesia, intensive care and pain therapy. Followed by digital storage for the finding.
  After the subsequent operation, the investigator determines whether knowledge of detected pathologies would have an effective influence on the anesthesiological procedure or not.

SUMMARY:
Introduction: The uncomplicated and focused transthoracic cardiac ultrasound examination, which is gentle for the patient, gives the doctor in a short time a lot of information about possible, as unrecognized pathologies of the organs of the chest.

Before a patient undergoes a planned procedure or intervention with a subsequent intensive stay, examinations are necessary from which the anesthetist/intensive physician has important information the state of health of the patient. The findings and the information will be used to plan the individual anesthesia procedures and intensive medical management, which is suitable for the patient.

The aim of this work is to investigate whether the use of a modified examination protocol in patients who need to be admitted to an intensive care unit has an influence on the actions of the intensive care physician. Does the information that is collected from the findings have a complementary influence in the planning of intensive care management? The Study objectives

Primary objectives:

What is the frequency with which pathological changes are detected?

Secondary objectives:

Do the additional findings have an influence on the intensive care procedure?

DETAILED DESCRIPTION:
At the end of the 1980s, a protocol for transthoracic cardiac ultrasound examination was established in order to get a quick overview of the structure and function of a patient's heart. Under the abbreviation "FATE" (focus assessed transthoracic echocardiography), it was "FAST"(focused assessment with sonography for trauma) when it was analogous to the ultrasound examination in traumatized patients, became an important component in the care of the acutely ill patients ( Walcher.F et al,2009).

The uncomplicated and focused transthoracic cardiac ultrasound examination, which is gentle for the patient, gives the doctor in a short time a lot of information about possible, as unrecognized pathologies of the organs of the chest.

In 2014, M.T. Bétker et al. published a study on the preoperative transthoracic sonography of the heart. Pathologies were detected in 27 percent of the patients included in the study, that could have a possible influence on the anesthesiological and intensive medical care procedures (Bøtker, M.T et al,2014).

The aim of this work is to investigate whether the use of a modified examination protocol in patients who need to be admitted to an intensive care unit has an influence on the actions of the intensive care physician. Does the information that is collected from the findings have a complementary influence in the planning of intensive care management? Before a patient undergoes a planned procedure or intervention with a subsequent intensive stay, examinations are necessary from which the anesthetist/intensive physician has important information the state of health of the patient. The findings and the information will be used to plan the individual anesthesia procedures and intensive medical management, which is suitable for the patient.

The examination takes place as part of the premedication visit. In addition to the history and the physical examination, the evaluation of already carried out examinations takes place here. Potential risks and complications are also discussed if the patient desires.

This evaluation helps to reduce the perioperative and interventional risks for the patient. particularly the detection of the cardiopulmonary capacity of the patient. Various technical studies can help to diagnose diseases of the heart, lungs and vascular system or to record the course of a known disorder (Anästh. Intensivmed (51) ,2010).

In addition to laboratory examinations, the electrocardiogram, the X-ray examination of the organs of the thorax, the blood vessel sonography, echocardiography is available.

The most common indications of echocardiography are the assessment of left and right ventricular pumping function and the exclusion of cardiac defects and shunt in patients with signs of heart failure or pathological auscultation findings.

These findings will be analyzed latest the day before a planned operation or intervention during the premedication visits and discussed with the patient in order to develop a patient-specific procedure and regimen.

This possibility exists for urgent interventions or interventions that which must be carried out on the same day, only conditionally and not for all planned admissions in the intensive care unit. Completeness of anesthetic and intensive medical findings about a statement the cardiopulmonary function is not always to be expected. In favor of rapid therapy, this must usually be dispensed with in a patient-individual risk-benefit-assessment.

The purpose of this study is to help answer the question whether the routine use of focused transthoracic echocardiography in unplanned admission to the Intensive Care Unit is a useful additional measure for the anesthesiologist and intensive physician in order to provide the patient with more safety?

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Age: greater than 60 years old
* Unplanned admission to the intensive care unit
* The patient's or caregiver's ability to educate
* Existing approval of the study

Exclusion Criteria:

* Lack of consent
* Alter < 60 years old
* • Non-Informable Patient.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Detection the pathological changes and finding of the Heart and the lung by using the Transesophgeal Echocardiography | It take over for every patient about 20 minutes to 30 minutes
  Using the Transesophgeal Echocardiography to detect the pathological changes and finding of the Heart and the lung (Percardial effusion in centimeter,pleural effusion in centimeter,ejection fraction in percentage,left ventricular hypertrophy in centimeter)

SECONDARY OUTCOMES:
Correlation between the finding that will be detected by transesophageal Echocardiography (TEE) and the management plan of the patient | from the first day of admission in the intensive care up to three days

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelsalam, Master, Principal Investigator — Vivantes Auguste-Viktoria-Klinikum
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No